CLINICAL TRIAL: NCT01375101
Title: Therapeutic Effect of Quercetin and the Current Treatment of Erosive and Atrophic Oral Lichen Planus
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Mashhad University of Medical Sciences (Other)
Responsible Party: maryam amirchaghmaghi, assistant professor of oral medicine department- mashhad medical school
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 88705
Record Dates: First submitted 2011-06-14; First posted 2011-06-17 (Estimated); Last update posted 2011-07-26 (Estimated); Status verified 2011-07

CONDITIONS: Atrophic Oral Lichen Planus; Erosive Oral Lichen Planus
Keywords: lichen planus; quercetin
MeSH Terms: conditions — Lichen Planus | interventions — Quercetin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor

ARMS (2):
- quercetin (Active Comparator): quercetin is one of flavonoids , and having therapeutical anti-inflammatory and antioxidant action
  Interventions: Drug: Quercetin
- placebo (Placebo Comparator): placebo capsul is produced with lactose for using in placebo/ control group.
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: placebo — The patient is directed to use placebo capsule two times a day, ,until the one mouth
  Arms: placebo
Drug: Quercetin — The patient is directed to digest quercetin hydrate capsule two times a day,until one mouth
  Arms: quercetin

SUMMARY:
Lichen planus (LP) is a common chronic inflammatory mucocutaneous disease with an immunologic etiology ,which has number of different clinical forms. Alternative natural or herbal origine drugs with antioxidant and anti-inflammatory properties have been used individually or in combination with systemic corticosteroids in order to decrease adverse drug reactions.

This study was conducted to evaluate the effect of quercetin on treatment of erosive -atrophic lesions of oral lichen planus (OLP).

ELIGIBILITY:
Inclusion Criteria:

* confirmation of clinical diagnosis of Atrophic and erosive lichen planus by histological examination
* two weeks wash out periods after the last treatment
* having the experience of atrophic and erosive lesion greater than 1 cm having the experience of pain and burning greater than 3.5 in VAS Score

Exclusion Criteria:

* confirmation of dysplasia and malignancy in histologic examination
* confirmation of lichenoid reaction in histologic examination
* pregnancy and breast feeding
* using fluorokinolon and cyclosporin which interact with quercetin

Ages: 12 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 30 (Estimated)
Dates: Start 2010-04; Primary Completion 2011-09 (Estimated); Study Completion 2011-09 (Estimated)

PRIMARY OUTCOMES:
the effects of this Drug on OLP measured with VAS scale for pain and evaluation of intensity of lesions. | 2 months
  In the present work the Analogical Visual Scale is used TO evaluate pain,and we also record the intensity of lesions weekly and any side effect of this Drug

CONTACTS AND LOCATIONS:
Locations (1):
- Mashhad university of Medical science, Research Center of oral and maxillofacial medicine, Mashhad, Khorasan Razavi, Iran